CLINICAL TRIAL: NCT05312801
Title: LMY-920 for Treatment of Relapsed or Refractory Non-Hodgkin Lymphoma
Brief Title: Phase 1 Study of BAFF CAR-T Cells (LMY-920) for Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Luminary Therapeutics (Industry)
Collaborators: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LMY-920-001
Record Dates: First submitted 2022-03-24; First posted 2022-04-06 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Lymphoma, Non-Hodgkin Lymphoma, B-Cell
Keywords: non-Hodgkin lymphoma.
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: Open label, dose escalation study.
  Dose Levels
  1. 1 x 10 million BAFF+ CAR cells/kg
  2. 2 x 10 million BAFF+ CAR cells/kg
  3. 4 x 10 million BAFF+ CAR cells/kg
  4. 8 x 10 million BAFF+ CAR cells/kg
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LMY-920 dose escalation (Experimental): Open label, dose escalation study with up to four dose levels of LMY-920. The maximum tolerated dose (MTD) of LMY-920 will be determined using dose-escalation 3+3 design.
  Interventions: Drug: BAFF CAR-T

INTERVENTIONS:
Drug: BAFF CAR-T — Autologous CAR-T cell therapy expressing the BAFF-ligand.
  Other Names: LMY-920

SUMMARY:
Therapy with chimeric antigen receptor T (CAR-T) cells has demonstrated activity against refractory lymphoma, however not all tumors respond or remain in response to CD19 targeted CAR-T cells. We posit that CAR-T cells expressing BAFF (BAFF CAR-T cells) can become another strategy to treat refractory lymphoma, even after relapse following cluster of differentiation antigen 19 (CD19) targeting CAR-T treatment.

This phase 1 study will evaluate safe dose and provide initial signal of the activity of BAFF CAR-T cells against relapsed non-Hodgkin lymphoma using a single lymphodepletion regimen and using a BAFF CAR-T cell manufacturing process.

DETAILED DESCRIPTION:
LMY-920 is an autologous CAR-T cell therapy consisting of autologous cluster of differentiation 4 (CD4) positive and cluster of differentiation 8 (CD8) positive human T cells that are genetically engineered using the non-viral transposon system to express the BAFF-ligand CAR-T that target BAFF receptor family members to eliminate malignant B cells.

BAFF receptor family includes B-cell activating factor receptor (BR3), B-cell maturation antigen (BCMA) and transmembrane activator and calcium modulator and cyclophilin ligand interactor (TACI). These receptors are present on non-Hodgkin lymphoma.

The goal of LMY-920-001 phase 1 study is to find recommended phase 2 dose of LMY-920 for treatment of patients with relapsed or refractory non-Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically confirmed non-Hodgkin lymphoma relapsed after 2 or more lines of therapy or disease refractory to chemotherapy (defined as progressive disease or stable disease lasting ≤6 months, as best response to most recent chemotherapy regimen; or disease progression or recurrence ≤12 months after prior autologous stem cell transplantation (ASCT).
2. No evidence of central nervous system (CNS) lymphoma.
3. Male or female > 18 years of age.
4. Eastern Cooperative Oncology Group Performance status ≤ 2.
5. At least one measurable lesion.
6. >2 weeks since prior radiation therapy or systemic therapy at the time of leukapheresis.
7. Total bilirubin ≤ 1.5 mg/dL (except in patients with Gilbert's syndrome).
8. Aspartate aminotransferase/alanine transferase ≤ 2.5 X institutional upper limit of normal.
9. Serum creatinine < 1.5 mg/dL.
10. Cardiac ejection fraction of >50%, and no evidence of pericardial effusion, as determined by an echocardiogram.
11. Adequate pulmonary function as defined as pulse oximetry ≥ 92% on room air.
12. Subjects (or legal guardians) must have the ability to understand and the willingness to sign a written informed consent document.
13. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 90 days after the BAFF CAR-T cell infusion.
14. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm.

Exclusion Criteria:

1. ASCT within 6 weeks of informed consent.
2. History of allogeneic hematopoietic stem cell transplantation.
3. Active graft-versus-host disease.
4. Active central nervous system or meningeal involvement by lymphoma or leukemia.
5. Active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast).
6. Less than 28 days elapsed between prior treatment with investigational agent(s) and the day of lymphocyte collection.
7. New York Heart Association class IV congestive heart failure.
8. Cardiovascular disorders including unstable angina pectoris, clinically significant cardiac arrhythmias, myocardial infarction or stroke (including transient ischemic attack, or other ischemic event) within 6 months prior to registration.
9. Active infection requiring intravenous systemic treatment.
10. HIV seropositivity.
11. Pregnant or breastfeeding women.
12. Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy.
13. Serologic status reflecting active hepatitis B or C infection.
14. Patients with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.
15. Subjects with uncontrolled intercurrent illness.
16. Known additional malignancies which require systemic treatment.
17. History of autoimmune disease with requirement of immunosuppressive medications (other than low dose steroids) within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
To determine recommended phase II dose of human LMY-920. | 24 months
  Maximum tolerated dose.

SECONDARY OUTCOMES:
To establish toxicity profile for the infusion of LMY-920. | 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. All adverse events during study will be collected, categorized, and graded. Attribution of relatedness to the investigational agent will be assigned.
To determine the objective response rate . | 24 months
  Response rate.
To determine the complete response rate. | 24 months
  Response rate.
To determine the duration of response. | 24 months
  Duration of response.
To determine the progression-free survival. | 24 months
  Progression-free survival.
To determine the overall survival. | 24 months
  Overall survival.
To determine incidence of adverse events. | 24 months
  Incidence of adverse events.
To determine incidence of anti- LMY-920 antibodies. | 24 months
  Incidence of anti- LMY-920 antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo F. Caimi, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute
Locations (2):
- United States (2):
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Taussig Cancer Institute | Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No